CLINICAL TRIAL: NCT00297115
Title: Effect of Roflumilast on Exacerbation Rate in Patients With COPD. The HERMES Study
Brief Title: Effect of Roflumilast on Exacerbation Rate in Patients With Chronic Obstructive Pulmonary Disease (COPD): The HERMES Study (BY217/M2-125)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY217/M2-125
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Results first posted 2011-05-19 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Roflumilast; COPD; Chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Roflumilast (Active Comparator): 500 mcg, once daily, oral administration in the morning
  Interventions: Drug: Roflumilast
- Placebo (Placebo Comparator): once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — 500 mcg, once daily, oral administration in the morning
  Arms: Roflumilast
Drug: Placebo — once daily
  Arms: Placebo

SUMMARY:
The aim of the study is to compare the effect of roflumilast on exacerbation rate and pulmonary function in patients with chronic obstructive pulmonary disease (COPD). Roflumilast will be administered orally once daily in the morning at one dose level. The study duration will be up to 56 weeks. The study will provide further data on safety and tolerability of roflumilast.

For additional information (for US patients only) see www.COPDSTUDY.net or dial 866-788-2673 (toll free).

ELIGIBILITY:
Main Inclusion Criteria:

* COPD patients having at least one exacerbation within last year
* FEV1/FVC ratio (post-bronchodilator) ≤ 70%
* FEV1 (post-bronchodilator) ≤ 50% of predicted

Main Exclusion Criteria:

* COPD exacerbation not resolved at first baseline visit
* Diagnosis of asthma and/or other relevant lung disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1568 (Actual)
Dates: Start 2006-03; Primary Completion 2008-04 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (249):
- United States (134):
  - Altana Pharma/Nycomed Investigational Site, Bayou La Batre, Alabama
  - Altana Pharma/Nycomed Investigational Site, Birmingham, Alabama
  - Altana Pharma/Nycomed Investigational Site, Huntsville, Alabama
  - Altana Pharma/Nycomed Investigational Site, Bullhead City, Arizona
  - Altana Pharma/Nycomed Investigational Site, Phoenix, Arizona
  - Altana Pharma/Nycomed Investigational Site, Fort Smith, Arkansas
  - Altana Pharma/Nycomed Investigational Site, Little Rock, Arkansas
  - Altana Pharma/Nycomed Investigational Site, Anaheim, California
  - Altana Pharma/Nycomed Investigational Site, Burbank, California
  - Altana Pharma/Nycomed Investigational Site, Carlsbad, California
  - Altana Pharma/Nycomed Investigational Site, Fresno, California
  - Altana Pharma/Nycomed Investigational Site, Lakewood, California
  - Altana Pharma/Nycomed Investigational Site, Long Beach, California
  - Altana Pharma/Nycomed Investigational Site, Los Alamitos, California
  - Altana Pharma/Nycomed Investigational Site, Los Angeles, California
  - Altana Pharma/Nycomed Investigational Site, Roseville, California
  - Altana Pharma/Nycomed Investigational Site, Sacramento, California
  - Altana Pharma/Nycomed Investigational Site, San Diego, California
  - Altana Pharma/Nycomed Investigational Site, Sepulveda, California
  - Altana Pharma/Nycomed Investigational Site, Stockton, California
  - Altana Pharma/Nycomed Investigational Site, Denver, Colorado
  - Altana Pharma/Nycomed Investigational Site, Waterbury, Connecticut
  - Altana Pharma/Nycomed Investigational Site, Washington D.C., District of Columbia
  - Altana Pharma/Nycomed Investigational Site, Clearwater, Florida
  - Altana Pharma/Nycomed Investigational Site, DeLand, Florida
  - Altana Pharma/Nycomed Investigational Site, Fort Lauderdale, Florida
  - Altana Pharma/Nycomed Investigational Site, Jacksonville, Florida
  - Altana Pharma/Nycomed Investigational Site, Miami, Florida
  - Altana Pharma/Nycomed Investigational Site, Miami Beach, Florida
  - Altana Pharma/Nycomed Investigational Site, Ocala, Florida
  - Altana Pharma/Nycomed Investigational Site, Ormand Beach, Florida
  - Altana Pharma/Nycomed Investigational Site, Port Orange, Florida
  - Altana Pharma/Nycomed Investigational Site, Tamarac, Florida
  - Altana Pharma/Nycomed Investigational Site, Vero Beach, Florida
  - Altana Pharma/Nycomed Investigational Site, Atlanta, Georgia
  - Altana Pharma/Nycomed Investigational Site, Blue Ridge, Georgia
  - Altana Pharma/Nycomed Investigational Site, Columbus, Georgia
  - Altana Pharma/Nycomed Investigational Site, Decatur, Georgia
  - Altana Pharma/Nycomed Investigational Site, Fort Eisenhower, Georgia
  - Altana Pharma/Nycomed Investigational Site, Marietta, Georgia
  - Altana Pharma/Nycomed Investigational Site, Rincon, Georgia
  - Altana Pharma/Nycomed Investigational Site, Savannah, Georgia
  - Altana Pharma/Nycomed Investigational Site, Twin Falls, Idaho
  - Altana Pharma/Nycomed Investigational Site, Champaign, Illinois
  - Altana Pharma/Nycomed Investigational Site, Chicago, Illinois
  - Altana Pharma/Nycomed Investigational Site, Elk Grove Village, Illinois
  - Altana Pharma/Nycomed Investigational Site, North Chicago, Illinois
  - Altana Pharma/Nycomed Investigational Site, Peoria, Illinois
  - Altana Pharma/Nycomed Investigational Site, River Forest, Illinois
  - Altana Pharma/Nycomed Investigational Site, Elkhart, Indiana
  - Altana Pharma/Nycomed Investigational Site, Indianapolis, Indiana
  - Altana Pharma/Nycomed Investigational Site, New Albany, Indiana
  - Altana Pharma/Nycomed Investigational Site, Dubuque, Iowa
  - Altana Pharma/Nycomed Investigational Site, Fort Dodge, Iowa
  - Altana Pharma/Nycomed Investigational Site, Iowa City, Iowa
  - Altana Pharma/Nycomed Investigational Site, Waterloo, Iowa
  - Altana Pharma/Nycomed Investigational Site, Olathe, Kansas
  - Altana Pharma/Nycomed Investigational Site, Topeka, Kansas
  - Altana Pharma/Nycomed Investigational Site, Campbellsville, Kentucky
  - Altana Pharma/Nycomed Investigational Site, Hazard, Kentucky
  - Altana Pharma/Nycomed Investigational Site, Louisville, Kentucky
  - Altana Pharma/Nycomed Investigational Site, Metairie, Louisiana
  - Altana Pharma/Nycomed Investigational Site, West Monroe, Louisiana
  - Altana Pharma/Nycomed Investigational Site, Columbia, Maryland
  - Altana Pharma/Nycomed Investigational Site, Boston, Massachusetts
  - Altana Pharma/Nycomed Investigational Site, Brighton, Michigan
  - Altana Pharma/Nycomed Investigational Site, Interlochen, Michigan
  - Altana Pharma/Nycomed Investigational Site, Livonia, Michigan
  - Altana Pharma/Nycomed Investigational Site, Portage, Michigan
  - Altana Pharma/Nycomed Investigational Site, Saginaw, Michigan
  - Altana Pharma/Nycomed Investigational Site, Duluth, Minnesota
  - Altana Pharma/Nycomed Investigational Site, Edina, Minnesota
  - Altana Pharma/Nycomed Investigational Site, Minneapolis, Minnesota
  - Altana Pharma/Nycomed Investigational Site, Rochester, Minnesota
  - Altana Pharma/Nycomed Investigational Site, Chesterfield, Missouri
  - Altana Pharma/Nycomed Investigational Site, Jefferson City, Missouri
  - Altana Pharma/Nycomed Investigational Site, Kansas City, Missouri
  - Altana Pharma/Nycomed Investigational Site, St Louis, Missouri
  - Altana Pharma/Nycomed Investigational Site, Sunset, Missouri
  - Altana Pharma/Nycomed Investigational Site, Bozeman, Montana
  - Altana Pharma/Nycomed Investigational Site, Butte, Montana
  - Altana Pharma/Nycomed Investigational Site, Omaha, Nebraska
  - Altana Pharma/Nycomed Investigational Site, Las Vegas, Nevada
  - Altana Pharma/Nycomed Investigational Site, Absecon, New Jersey
  - Altana Pharma/Nycomed Investigational Site, Hamilton, New Jersey
  - Altana Pharma/Nycomed Investigational Site, South Bound Brook, New Jersey
  - Altana Pharma/Nycomed Investigational Site, Camillus, New York
  - Altana Pharma/Nycomed Investigational Site, Corning, New York
  - Altana Pharma/Nycomed Investigational Site, Cortland, New York
  - Altana Pharma/Nycomed Investigational Site, New Hyde Park, New York
  - Altana Pharma/Nycomed Investigational Site, Syracuse, New York
  - Altana Pharma/Nycomed Investigational Site, Charlotte, North Carolina
  - Altana Pharma/Nycomed Investigational Site, Huntersville, North Carolina
  - Altana Pharma/Nycomed Investigational Site, Winston-Salem, North Carolina
  - Altana Pharma/Nycomed Investigational Site, Canton, Ohio
  - Altana Pharma/Nycomed Investigational Site, Cincinnati, Ohio
  - Altana Pharma/Nycomed Investigational Site, Columbus, Ohio
  - Altana Pharma/Nycomed Investigational Site, Sylvania, Ohio
  - Altana Pharma/Nycomed Investigational Site, Toledo, Ohio
  - Altana Pharma/Nycomed Investigational Site, Oklahoma City, Oklahoma
  - Altana Pharma/Nycomed Investigational Site, Medford, Oregon
  - Altana Pharma/Nycomed Investigational Site, Portland, Oregon
  - Altana Pharma/Nycomed Investigational Site, Erie, Pennsylvania
  - Altana Pharma/Nycomed Investigational Site, Hershey, Pennsylvania
  - Altana Pharma/Nycomed Investigational Site, Philadelphia, Pennsylvania
  - Altana Pharma/Nycomed Investigational Site, Pittsburgh, Pennsylvania
  - Altana Pharma/Nycomed Investigational Site, Stoneboro, Pennsylvania
  - Altana Pharma/Nycomed Investigational Site, Swarthmore, Pennsylvania
  - Altana Pharma/Nycomed Investigational Site, Johnston, Rhode Island
  - Altana Pharma/Nycomed Investigational Site, Charleston, South Carolina
  - Altana Pharma/Nycomed Investigational Site, Greenville, South Carolina
  - Altana Pharma/Nycomed Investigational Site, Greer, South Carolina
  - Altana Pharma/Nycomed Investigational Site, Union, South Carolina
  - Altana Pharma/Nycomed Investigational Site, Williamston, South Carolina
  - Altana Pharma/Nycomed Investigational Site, Johnson City, Tennessee
  - Altana Pharma/Nycomed Investigational Site, Knoxville, Tennessee
  - Altana Pharma/Nycomed Investigational Site, Memphis, Tennessee
  - Altana Pharma/Nycomed Investigational Site, Nashville, Tennessee
  - Altana Pharma/Nycomed Investigational Site, New Tazewell, Tennessee
  - Altana Pharma/Nycomed Investigational Site, Boerne, Texas
  - Altana Pharma/Nycomed Investigational Site, Corsicana, Texas
  - Altana Pharma/Nycomed Investigational Site, Fort Worth, Texas
  - Altana Pharma/Nycomed Investigational Site, Houston, Texas
  - Altana Pharma/Nycomed Investigational Site, Hurst, Texas
  - Altana Pharma/Nycomed Investigational Site, McKinney, Texas
  - Altana Pharma/Nycomed Investigational Site, San Antonio, Texas
  - Altana Pharma/Nycomed Investigational Site, Seguin, Texas
  - Altana Pharma/Nycomed Investigational Site, Tyler, Texas
  - Altana Pharma/Nycomed Investigational Site, Salt Lake City, Utah
  - Altana Pharma/Nycomed Investigational Site, Lynchburg, Virginia
  - Altana Pharma/Nycomed Investigational Site, Seattle, Washington
  - Altana Pharma/Nycomed Investigational Site, Spokane, Washington
  - Altana Pharma/Nycomed Investigational Site, Charleston, West Virginia
  - Altana Pharma/Nycomed Investigational Site, Glendale, Wisconsin
- Canada (38):
  - Altana Pharma/Nycomed Investigational Site, Calgary, Alberta
  - Altana Pharma/Nycomed Investigational Site, Edmonton, Alberta
  - Altana Pharma/Nycomed Investigational Site, Spruce Grove, Alberta
  - Altana Pharma/Nycomed Investigational Site, Burnaby, British Columbia
  - Altana Pharma/Nycomed Investigational Site, Penticton, British Columbia
  - Altana Pharma/Nycomed Investigational Site, Vancouver, British Columbia
  - Altana Pharma/Nycomed Investigational Site, Truro, Nova Scotia
  - Altana Pharma/Nycomed Investigational Site, Chatham, Ontario
  - Altana Pharma/Nycomed Investigational Site, Hamilton, Ontario
  - Altana Pharma/Nycomed Investigational Site, London, Ontario
  - Altana Pharma/Nycomed Investigational Site, Mississauga, Ontario
  - Altana Pharma/Nycomed Investigational Site, Ottawa, Ontario
  - Altana Pharma/Nycomed Investigational Site, Sarnia, Ontario
  - Altana Pharma/Nycomed Investigational Site, Scarborough Village, Ontario
  - Altana Pharma/Nycomed Investigational Site, Toronto, Ontario
  - Altana Pharma/Nycomed Investigational Site, Montreal, Quebec
  - Altana Pharma/Nycomed Investigational Site, Saint Romuald, Quebec
  - Altana Pharma/Nycomed Investigational Site, Sainte-Foy, Quebec
  - Altana Pharma/Nycomed Investigational Site, Sherbrooke, Quebec
  - Altana Pharma/Nycomed Investigational Site, Ste-Foy, Quebec
  - Altana Pharma/Nycomed Investigational Site, Antigonish
  - Altana Pharma/Nycomed Investigational Site, Bridgewater
  - Altana Pharma/Nycomed Investigational Site, Calgary
  - Altana Pharma/Nycomed Investigational Site, Corunna
  - Altana Pharma/Nycomed Investigational Site, Edmonton
  - Altana Pharma/Nycomed Investigational Site, Fort Erie
  - Altana Pharma/Nycomed Investigational Site, Grimsby
  - Altana Pharma/Nycomed Investigational Site, Hamilton
  - Altana Pharma/Nycomed Investigational Site, Longueuil
  - Altana Pharma/Nycomed Investigational Site, Montreal
  - Altana Pharma/Nycomed Investigational Site, Ontario
  - Altana Pharma/Nycomed Investigational Site, Richmond Hill
  - Altana Pharma/Nycomed Investigational Site, Saint John
  - Altana Pharma/Nycomed Investigational Site, Saint-Jérôme
  - Altana Pharma/Nycomed Investigational Site, Saint-Léonard
  - Altana Pharma/Nycomed Investigational Site, Sherbrooke
  - Altana Pharma/Nycomed Investigational Site, Toronto
  - Altana Pharma/Nycomed Investigational Site, Winnipeg
- Germany (12):
  - Altana Pharma/Nycomed Investigational Site, Berlin
  - Altana Pharma/Nycomed Investigational Site, Donaustauf
  - Altana Pharma/Nycomed Investigational Site, Großhansdorf
  - Altana Pharma/Nycomed Investigational Site, Halle
  - Altana Pharma/Nycomed Investigational Site, Hamburg
  - Altana Pharma/Nycomed Investigational Site, Landsberg/Lech
  - Altana Pharma/Nycomed Investigational Site, Neuruppin
  - Altana Pharma/Nycomed Investigational Site, Oschersleben
  - Altana Pharma/Nycomed Investigational Site, Potsdam
  - Altana Pharma/Nycomed Investigational Site, Regensburg
  - Altana Pharma/Nycomed Investigational Site, Rüdersdorf
  - Altana Pharma/Nycomed Investigational Site, Ulm
- India (16):
  - Altana Pharma/Nycomed Investigational Site, Bangalore
  - Altana Pharma/Nycomed Investigational Site, Bangalore, Karnataka
  - Altana Pharma/Nycomed Investigational Site, Chennai
  - Altana Pharma/Nycomed Investigational Site, Coimbatore
  - Altana Pharma/Nycomed Investigational Site, Coimbatore, Tamilnadu
  - Altana Pharma/Nycomed Investigational Site, Goa
  - Altana Pharma/Nycomed Investigational Site, Hyderabad
  - Altana Pharma/Nycomed Investigational Site, Indore, South Tukuganj
  - Altana Pharma/Nycomed Investigational Site, Mangalore
  - Altana Pharma/Nycomed Investigational Site, Mumbai
  - Altana Pharma/Nycomed Investigational Site, Mumbai, Byculla
  - Altana Pharma/Nycomed Investigational Site, Mumbai, Dadar (E)
  - Altana Pharma/Nycomed Investigational Site, Mysore
  - Altana Pharma/Nycomed Investigational Site, Nagpur
  - Altana Pharma/Nycomed Investigational Site, Pune
  - Altana Pharma/Nycomed Investigational Site, Shastri Nagar, Jaipur
- Italy (11):
  - Altana Pharma/Nycomed Investigational Site, Bergamo
  - Altana Pharma/Nycomed Investigational Site, Bologna
  - Altana Pharma/Nycomed Investigational Site, Cassano Murge
  - Altana Pharma/Nycomed Investigational Site, Florence
  - Altana Pharma/Nycomed Investigational Site, Milan
  - Altana Pharma/Nycomed Investigational Site, Parma
  - Altana Pharma/Nycomed Investigational Site, Pavia
  - Altana Pharma/Nycomed Investigational Site, Roma
  - Altana Pharma/Nycomed Investigational Site, Trieste
  - Altana Pharma/Nycomed Investigational Site, Verona
  - Altana Pharma/Nycomed Investigational Site, Veruno
- Poland (10):
  - Altana Pharma/Nycomed Investigational Site, Chrzanów
  - Altana Pharma/Nycomed Investigational Site, Częstochowa
  - Altana Pharma/Nycomed Investigational Site, Działdowo
  - Altana Pharma/Nycomed Investigational Site, Katowice
  - Altana Pharma/Nycomed Investigational Site, Krakow
  - Altana Pharma/Nycomed Investigational Site, Lublin
  - Altana Pharma/Nycomed Investigational Site, Poznan
  - Altana Pharma/Nycomed Investigational Site, Warsaw
  - Altana Pharma/Nycomed Investigational Site, Wodzisław Śląski
  - Altana Pharma/Nycomed Investigational Site, Zgierz
- South Africa (12):
  - Altana Pharma/Nycomed Investigational Site, Bellville, Cape Town
  - Altana Pharma/Nycomed Investigational Site, Berea, Durban
  - Altana Pharma/Nycomed Investigational Site, Bloemfontein
  - Altana Pharma/Nycomed Investigational Site, C/O Netcare & Garsfontein Roads
  - Altana Pharma/Nycomed Investigational Site, Cape Town
  - Altana Pharma/Nycomed Investigational Site, Cape Town, Tygerberg
  - Altana Pharma/Nycomed Investigational Site, Durban, Amanzimtoti
  - Altana Pharma/Nycomed Investigational Site, Durbanville / Cape Town
  - Altana Pharma/Nycomed Investigational Site, Mowbray, Cape Town
  - Altana Pharma/Nycomed Investigational Site, Paarl, Cape Town
  - Altana Pharma/Nycomed Investigational Site, Pretoria
  - Altana Pharma/Nycomed Investigational Site, Somerset West
- Spain (16):
  - Altana Pharma/Nycomed Investigational Site, Badajoz
  - Altana Pharma/Nycomed Investigational Site, Calde (Lugo)
  - Altana Pharma/Nycomed Investigational Site, Cartagena
  - Altana Pharma/Nycomed Investigational Site, Elda
  - Altana Pharma/Nycomed Investigational Site, Getafe
  - Altana Pharma/Nycomed Investigational Site, Guadalajara
  - Altana Pharma/Nycomed Investigational Site, Madrid
  - Altana Pharma/Nycomed Investigational Site, Merida (Badajoz)
  - Altana Pharma/Nycomed Investigational Site, Partida de Bacarot (Alicante)
  - Altana Pharma/Nycomed Investigational Site, Pontevedra
  - Altana Pharma/Nycomed Investigational Site, Requena
  - Altana Pharma/Nycomed Investigational Site, Santiago de Compostela
  - Altana Pharma/Nycomed Investigational Site, Talavera de La Reina (Toledo)
  - Altana Pharma/Nycomed Investigational Site, Tarrasa (Barcelona)
  - Altana Pharma/Nycomed Investigational Site, Toldeo
  - Altana Pharma/Nycomed Investigational Site, Valencia

REFERENCES:
- [Result] Calverley PM, Rabe KF, Goehring UM, Kristiansen S, Fabbri LM, Martinez FJ; M2-124 and M2-125 study groups. Roflumilast in symptomatic chronic obstructive pulmonary disease: two randomised clinical trials. Lancet. 2009 Aug 29;374(9691):685-94. doi: 10.1016/S0140-6736(09)61255-1. PMID 19716960
- [Derived] Facius A, Krause A, Claret L, Bruno R, Lahu G. Modeling and Simulation of Pivotal Clinical Trials Using Linked Models for Multiple Endpoints in Chronic Obstructive Pulmonary Disease With Roflumilast. J Clin Pharmacol. 2017 Aug;57(8):1042-1052. doi: 10.1002/jcph.885. Epub 2017 Apr 17. PMID 28419462
- [Derived] Hanania NA, Calverley PM, Dransfield MT, Karpel JP, Brose M, Zhu H, Goehring UM, Rowe P. Pooled subpopulation analyses of the effects of roflumilast on exacerbations and lung function in COPD. Respir Med. 2014 Feb;108(2):366-75. doi: 10.1016/j.rmed.2013.09.018. Epub 2013 Sep 30. PMID 24120253
- [Derived] Wedzicha JA, Rabe KF, Martinez FJ, Bredenbroker D, Brose M, Goehring UM, Calverley PMA. Efficacy of roflumilast in the COPD frequent exacerbator phenotype. Chest. 2013 May;143(5):1302-1311. doi: 10.1378/chest.12-1489. PMID 23117188
- [Derived] Cazzola M, Picciolo S, Matera MG. Roflumilast in chronic obstructive pulmonary disease: evidence from large trials. Expert Opin Pharmacother. 2010 Feb;11(3):441-9. doi: 10.1517/14656560903555201. PMID 20102307

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Roflumilast | Placebo
Started | 772 (Includes all randomized patients who took at least one dose of the investigational drug.) | 796 (Includes all randomized patients who took at least one dose of the investigational drug.)
Completed | 527 | 550
Not Completed | 245 | 246

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast | Placebo | Total
Number analyzed (Participants) | 772 | 796 | 1568
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.92 (9.2) | 64.31 (9.0) | 64.12 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 148 | 310
  Male | 610 | 648 | 1258

OUTCOME MEASURES:

1. Primary Outcome: Pre-bronchodilator Forced Expiratory Volume in First Second (FEV1)
Description: Mean change from baseline during the treatment period in pre-bronchodilator FEV1 [L]
Time Frame: Change from baseline over 52 weeks of treatment
Population: ITT (Intention to Treat) analysis. Number of participants analyzed = number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 730 | 766
mL | 33 (7) | -25 (7)
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment of the significance level was done as a hierarchical approach for hypotheses testing was used; Repeated measurements analysis (change from baseline over 52 weeks of treatment taking all post-randomization measurements into account); Mean Difference (Net) = 58, 95% CI 2-sided [41 to 75], Standard Error of Mean 9

2. Primary Outcome: COPD Exacerbation Rate (Moderate or Severe)
Description: Mean rate of COPD exacerbations requiring oral or parenteral glucocorticosteroids (=moderate COPD exacerbations), or requiring hospitalization, or leading to death (=severe COPD exacerbations), per patient per year. A COPD exacerbation is an event in the natural course of the disease characterized by a change in the patient's baseline dyspnea, cough and/or sputum beyond day-to-day variability sufficient to warrant a change in management [American Thoracic Society (ATS) / European Respiratory Society (ERS) 2005].
Time Frame: 52 weeks treatment period
Population: ITT analysis.
Measure: Mean (95% Confidence Interval); unit: exacerbations per patient per year
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 772 | 796
exacerbations per patient per year | 1.210 [1.074 to 1.364] | 1.485 [1.333 to 1.655]
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p = 0.0035, Poisson regression — No adjustment of the significance level was done as a hierarchical approach for hypotheses testing was used; Rate ratio = 0.815, 95% CI 2-sided [0.710 to 0.935], Standard Error of Mean 0.057

3. Secondary Outcome: Post-bronchodilator FEV1 [L]
Description: Mean change from baseline during the treatment period in post-bronchodilator FEV1 [L]
Time Frame: Change from baseline over 52 weeks of treatment
Population: ITT analysis. Number of participants analyzed = number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 724 | 764
mL | 44 (7) | -17 (7)
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment of the significance level was done as a hierarchical approach for hypotheses testing was used; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 61, 95% CI 2-sided [44 to 79], Standard Error of Mean 9

4. Secondary Outcome: Time to Mortality Due to Any Reason
Time Frame: 52 weeks treatment period
Population: ITT analysis. Number of participants analyzed = number of participants who died.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 25 | 25
days | 201.0 (116.9) | 214.6 (137.3)
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p = 0.5028, Cox proportional hazards regression — No adjustment of the significance level was done as a hierarchical approach for hypotheses testing was used; Hazard Ratio (HR) = 1.213, 95% CI 2-sided [0.689 to 2.137], Standard Error of Mean 0.350 — The statistical analysis is based on the ITT Analysis Set (n= 772 in the roflumilast group, n= 796 in the placebo group)

5. Secondary Outcome: Natural Log-transformed C-reactive Protein (CRP)
Description: Mean change from baseline to the last post randomization measurement in natural log-transformed CRP
Time Frame: Change from baseline to last post randomization measurement (52 weeks)
Population: ITT analysis. Number of participants analyzed = number of participants with data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 680 | 696
mg/L | 1.0840 [0.9766 to 1.2033] | 1.0233 [0.9228 to 1.1348]
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p = 0.3627, ANCOVA — No adjustment of the significance level was done as a hierarchical approach for hypotheses testing was used; ANCOVA model including last observation carried forward (LOCF) method; Mean Difference calculated as ratio = 1.0593, 95% CI 2-sided [0.9356 to 1.1994]

6. Secondary Outcome: Mean Transition Dyspnea Index (TDI) Focal Score During the Treatment Period
Description: The TDI is a recognized questionnaire to measure dyspnea in an out patient COPD population. At baseline, 3 components of dyspnea, each graded with 4 questions, were asked: - Functional Impairment - Magnitude of Task - Magnitude of Effort At each of the post-randomization visits questions from the TDI were asked related to 3 components: Change in - Functional Impairment - Magnitude of Task - Magnitude of Effort Each question in the TDI is graded from -3 (major deterioration) to +3 (major improvement). This results in a TDI Focal Score ranging from -9 to +9.
Time Frame: Change from baseline over 52 weeks of treatment
Population: ITT analysis. Number of participants analyzed = number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 729 | 769
scores on a scale | 0.662 (0.087) | 0.376 (0.084)
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p = 0.0059, ANCOVA — No adjustment of the significance level was done as a hierarchical approach for hypotheses testing was used; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.286, 95% CI 2-sided [0.082 to 0.489], Standard Error of Mean 0.104

ADVERSE EVENTS:
Time Frame: 52 weeks treatment period
Description: The Safety Set was based on all randomized patients who took at least one dose of the investigational drug after randomization. Six patients randomized to placebo received roflumilast instead and were included in the roflumilast group for safety analyses.
Arm/Group | Roflumilast | Placebo
Serious Adverse Events (participants affected / at risk) | 157/778 | 183/790
Other Adverse Events (participants affected / at risk) | 145/778 | 81/790
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roflumilast (N=778) | Placebo (N=790)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 87 (110) | 121 (160)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (6)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 18 (18) | 10 (10)
Bronchopneumonia (Infections and infestations) | 1 (1) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia primary atypical (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 4 (4)
Angina pectoris (Cardiac disorders) | 2 (2) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 3 (3) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 3 (3)
Right ventricular failure (Cardiac disorders) | 1 (1) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (3)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cor pulmonale (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 2 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour of the small bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 2 (2) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 3 (3)
Chest pain (General disorders) | 0 (0) | 3 (3)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Death (General disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Metaplasia (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Ulcer haemorrhage (General disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 3 (3)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Anoxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Wernicke's encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Device dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye penetration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body trauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arterial stenosis (Vascular disorders) | 0 (0) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 3 (3) | 1 (1)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Endarterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (2) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roflumilast (N=778) | Placebo (N=790)
Diarrhoea (Gastrointestinal disorders) | 64 (71) | 23 (25) — non-serious
Weight decreased (Investigations) | 65 (67) | 20 (20)
Nasopharyngitis (Infections and infestations) | 35 (43) | 47 (57)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study results may be published and/or presented at scientific meetings. Prior to any submission, all manuscripts/abstracts must be presented to the sponsor for possible comments.